CLINICAL TRIAL: NCT05976581
Title: Using Probability of Community-Acquired Pneumonia to Tailor Antimicrobials Among Inpatients
Acronym: UP-CAPTAIn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Baghdadi (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jonathan Baghdadi, Assistant Professor, University of Maryland, Baltimore
Organization: University of Maryland, Baltimore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00103497
Record Dates: First submitted 2023-07-11; First posted 2023-08-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pneumonia; Pneumonia, Viral; Pneumonia, Bacterial
Keywords: diagnostic stewardship; antimicrobial stewardship
MeSH Terms: conditions — Pneumonia; Pneumonia, Viral; Pneumonia, Bacterial

STUDY DESIGN:
Intervention Model Description: This study involves a randomized trial embedded within a quasi-experiment. During the 1-year study period, we anticipate that 1,500 patients will be exposed to the electronic health record modification performed as part of the quasi-experiment. Regarding the randomized trial, if 100 patients are enrolled during the 1-year study period, including 50 in intervention patients and 50 controls, we anticipate that we will have sufficient precision to estimate the difference in binary outcomes (e.g., antibiotic discontinuation within 5 days) between the two groups with a margin of error of approximately 15% based on a 95% confidence interval.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electronic alert plus structured communication of test results (Experimental): An electronic health record alert will guide diagnostic testing for pneumonia. For patients with low or moderate probability of bacterial pneumonia, test results will be communicated to the primary team with guidance to consider discontinuing or de-escalating antibiotics.
  Interventions: Behavioral: Electronic alert; Behavioral: Structured communication of test results
- Electronic alert without structured communication of test results (Active Comparator): An electronic health record alert will guide diagnostic testing for pneumonia. The primary care team will access and interpret test results and decide upon composition and duration of antimicrobial without external guidance.
  Interventions: Behavioral: Electronic alert

INTERVENTIONS:
Behavioral: Electronic alert — An alert will appear in the electronic health record that provides options for diagnostic testing based on low, medium, or high probability of bacterial pneumonia.
Behavioral: Structured communication of test results — A clinical research team member will send an electronic message to the primary care team on behalf of the antimicrobial stewardship program with structured guidance to stop or de-escalate antibiotics and document these recommendations in the patient's chart.
  Arms: Electronic alert plus structured communication of test results

SUMMARY:
The goal of this prospective randomized study is to improve antibiotic use among hospitalized patients with suspected pneumonia. An alert was built into the electronic health record to guide use of diagnostic testing based on probability of bacterial pneumonia. Patients with test results suggesting viral infection will be randomized to either: (1) receive a structured communication from the antimicrobial stewardship team to de-escalate antibiotics or (2) usual care.

DETAILED DESCRIPTION:
Low-risk patients with viral pneumonia do not benefit from and may be harmed by antibiotic therapy. In this study, an alert will appear in the electronic health record of patients undergoing molecular diagnostic testing for respiratory symptoms that provides options for diagnostic testing based on pre-test probability of bacterial infection. Patients with test results suggesting possible viral infection will be randomized to either usual care or to receive test results along with structured guidance from antimicrobial stewardship to consider discontinuing or de-escalating antibiotics. This guidance, which will include an explicit calculation of the post-test probability of bacterial infection based on considering risk factors, vital signs, symptoms, and available imaging, will be communicated to the primary care team via direct electronic message and a summary note in the patient's chart. The final decision on whether to continue antibiotic therapy will be up to the primary team. The primary outcome of interest will be in-hospital antibiotic use. Safety outcomes will include length of stay, readmissions, hospital-free days, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the University of Maryland Medical Center or University of Maryland Medical Center-Midtown Campus who are prescribed antibiotics for suspected community-acquired respiratory infection.
* Protocol-based diagnostic testing supports possible viral infection, either by positive molecular test or low procalcitonin value.

Exclusion Criteria:

* Hospitalization for >72 hours prior to protocol-based diagnostic testing.
* Previous molecular testing for viral infection during the same hospital encounter.
* Severely immunosuppressed, defined as having hematologic malignancy, solid organ tumor on chemotherapy, or solid organ transplant on immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Hospital antibiotic days of therapy | Up to 90 days after randomization
  The aggregate sum of days for which any amount of a specific antimicrobial agent was administered during the hospital encounter, from arrival in the emergency department or on the hospital ward until discharge.

SECONDARY OUTCOMES:
Hospital length of stay | Up to 90 days after randomization
  Duration of hospitalization from admission to discharge
In-hospital mortality | Up to 90 days after randomization
  Death or discharge to hospice during initial hospitalization for any cause
Readmissions within 30-days of randomization | Within 30 days after randomization
  Readmissions for any cause within 30-days of randomization
C. difficile infections in the 30-days post-randomization | Within 30 days after randomization
  Positive test for C. difficile associated with initiation of antibiotics targeting C. difficile.
Acute kidney injury | Within 14 days of randomization
  Defined by an elevation in creatinine of > 0.5mg/dl or 2x baseline in a patient without previous end-stage renal disease.
Ventilator-free days in the 30-days post-randomization | 30 days after randomization.
  Days without a requirement for mechanical ventilation in the 30 days after randomization.
Hospital-free days in the 30-days post-randomization | 30 days after randomization.
  Days without hospitalization in the 30 days after randomization.
Antibiotic de-escalations within 72 hours after initiation | 3 days after randomization.
  Including narrowing, discontinuing, or converting the route of administration from intravenous to oral.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Morgan, MD, MS, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland Medical Center - Midtown Campus, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No